CLINICAL TRIAL: NCT06880029
Title: Circadian Rhythm Impact on Triple Negative Breast Cancer Response to Neoadjuvant Immunotherapy - a Feasibility Randomized Trial
Brief Title: Circadian Rhythm Impact on TNBC Response to Neoadjuvant Immunotherapy
Acronym: CIRCADIAN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government)
Responsible Party: Principal Investigator, Alexandra Guedes, Medical Oncologist Resident, Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 143/2024
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: TNBC; Immunotherapy; Circadian rhythm
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning Group (Experimental): All three neoadjuvant pembrolizumab cycles in the morning (before noon)
  Interventions: Other: Morning pembrolizumab infusions
- Afternoon Group (No Intervention): All three neoadjuvant pembrolizumab cycles in the afternoon (after noon)

INTERVENTIONS:
Other: Morning pembrolizumab infusions — Patients will be randomized 1:1 to receive all three neoadjuvant pembrolizumab cycles in the morning (before noon) or in the afternoon (after noon).
  Arms: Morning Group

SUMMARY:
CIRCADIAN is a prospective randomized clinical trial designed to evaluate the impact of pembrolizumab infusions' time-of-day on pathological complete response (pCR) rate among TNBC patients undergoing neoadjuvant treatment.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to receive all neoadjuvant pembrolizumab cycles (400 mg every 6 weeks) before versus after noon. Subjects will be stratified based on clinical stage at diagnosis (St. II vs III).

Primary outcome will be pCR rate. As a secondary outcome, we will assess for treatment related toxicity.

For planned exploratory circadian rhythm evaluation, daily body temperature and salivary cortisol variation will be measured before each ICI infusion and the Munich Chronotype Questionnaire (MCTQ) will be applied. To assess for emotional stress, physical exercise habits, stimulating substances use and light exposure, patients will also be subjected to the Distress Thermometer and a lifestyle questionnaire. For planned exploratory biomarker research, tumor infiltrating lymphocytes (TILs) analysis will be performed on the initial diagnostic biopsy and after surgery, on residual tumor (in patients not achieving pCR). Cytokine quantification and bulk RNA sequencing plus flow cytometry studies for immune populations profiling will be performed on peripheral blood, at baseline and before surgery, to check for potential biomarkers of circadian modulation.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 18 - 75 years old
* Diagnosed with Stage II or III TNBC and candidates for neoadjuvant treatment with ChT+pembrolizumab after multidisciplinary group discussion.

Exclusion Criteria:

* Patients unable to understand or consent to the study;
* Patients not completing ≥2 cycles of planned neoadjuvant pembrolizumab cycles or ≥50% of planned neoadjuvant ChT cycles;
* Patients under daily ≥10 mg of prednisolone or equivalent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | At the time of definitive surgery.
  Defined as ypT0/Tis ypN0, assessed by the local pathologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Região, Portugal